CLINICAL TRIAL: NCT02672761
Title: MBSR Improves Memory and Attention Due to a Stress Reduction as Opposed to Specific Memory Training
Brief Title: Effect of 8 Weeks of MBSR Training on Neuroplasticity and Improvement of Attention, Memory and Well-Being
Acronym: MBSR2015
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Thomas Frietsch, Prof. T. Frietsch, PhD, MD, MBA, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBSR-Diako-MA-2015
Record Dates: First submitted 2016-01-14; First posted 2016-02-03 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Stress
MeSH Terms: interventions — Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MBSR (Experimental): Subjects enrol and complete a standardized and licensed meditation program developed by Jon Kabat-Zinn. The program includes a weekly 200 min group session, daily meditation training from 20-40 min and one 4 h retreat within the study period. The individual daily and overall training volume is noted in min.
  Interventions: Behavioral: MBSR meditation
- MBT (Experimental): Subjects while being on the waiting list for MBSR are allocated to a web-based training program (MBT- My Brain Training) for working, episodic and general memory functions. The individual daily and overall training volume is noted in min.
  Interventions: Behavioral: MBT training
- Wellness (Active Comparator): Subjects while being on the waiting list for MBSR are allocated to a free accessable wellness program including sessions in a computerized chair delivering Shiatzu massage and relaxation music. The individual daily and overall training volume is noted in min.
  Interventions: Behavioral: Wellness
- Control (Placebo Comparator): Subjects while being on the waiting list for MBSR are requested to do no special program for stress reduction or memory improvement. The individual daily and overall training volume of sports or recreational activity is noted in min.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: MBSR meditation — Adopted from buddhism for western societies by Jon Kabat-Zinn, MBSR has been described as "a group program that focuses upon the progressive acquisition of mindful awareness, of mindfulness". The MBSR program is an eight-week workshop taught by certified trainers that entails weekly group meetings, homework, and instruction in three formal techniques: sitting mindfulness meditation, body scanning and simple yoga postures. Sitting meditation includes concentration on the breathing while not adhering to the flow of thoughts or emotions as well as the development of empathy and loving kindness for all persons. Body scanning is the first prolonged formal mindfulness technique taught during the first four weeks of the workshop, and entails quietly lying on one's back and focusing one's attention on various regions of the body, starting with the toes and moving up slowly to the top of the head.
  Arms: MBSR
Behavioral: MBT training — A specific memory brain training stimulates by a validated program according to Kawashima from the Industry University Research Project the according areas in the prefrontal lobe for calculation, logical reflection, optic/episodes and memory. The computerized program adopts to the difficulty level of the trainee. Selected were trainings for the categories "working/semantic" and "episodic/optical" memory and "logic/calculation" adjusted to the individual's selection from all categories but various themes (like sports, cars etc.).
  Arms: MBT
Behavioral: Wellness — The Brain Light Wellness chair is assessed for the stress reduction in industry and public Enterprises. In a European study 97% of subjects reported a stress reduction, improved well-being, performance and increased vitality, less fatigue and petulance. The chair "3D-Float-plus" system comprises of a massage chair in sitting to lying position, a headset with earphones a lighted glasses for visual and audio Stimulation. One standardized session of 45 min duration was chosen for the study that combined a short massage period with a relaxation trance session.
  Arms: Wellness
Behavioral: Control — The waiting period for the MBSR training to start simply should include no changes in lifestyle, recreational activity or intellectual training
  Arms: Control

SUMMARY:
Meditation improves attention and memory by reducing of the increased electric brain activity induced by a high stress level. This is associated to neuroplastic changes (volume reduction and/or neuron's density increases) in various brain structures. The question evolves if memory improvement by a standardized meditation program of 8 weeks (Mindfulness Based Stress Reduction MBSR) or a specific memory training (My Brain Training MBT) is a specific effect on brain networking or mediated by a reduced general activity induced by stress reduction. Thus, meditation or memory training should have differing neuroplastic effects.

The effects of memory function improvement by the respective training will be measured by MAT, a specific and validated computerized memory and attention test. Brain morphology is investigated by voxel based morphometry NMR before and immediately after an 8 weeks intervention period. Stress levels are measured by cortisol profiles of subjects. Compared were 4 groups- "MBSR" group- MBSR students after completed training, passive "control" group- subjects following an 8 weeks waiting period for the MBSR training without any memory training, active control "MBT" group- subjects on an 8 weeks waiting period for the MBSR training doing an 8 weeks MBT memory training instead, "Wellness" group - doing a structured program using relaxing massage and calming computerized chair ("Brain Light").

The hypothesis of the study is that MBSR improves memory function better than MBT when measured by MAT. Compared to both active and passive controls, MBSR training induces specific morphologic changes in the brain, indicated by a volume change of the voxel based morphometry method of 5% of a defined brain region. In comparison to smaller and less neuroplasticity induced by MBT on memory brain regions, MBSR induces greater volume changes on hippocampus and amygdala and stress reduction than the wellness program.

DETAILED DESCRIPTION:
The question evolves if memory improvement by a standardized meditation program of 8 weeks (Mindfulness Based Stress Reduction MBSR) or a specific memory training (My Brain Training MBT) is a specific effect on brain networking or mediated by a reduced general activity induced by stress reduction. The capacity of MBSR to induce dramatic neuroplastic changes such as morphological grey matter changes in the brain, reduced amygdala function and volume as well as electric activity level of the somatosensory cortex should allow for a discrimination and allocation of various memorial subfunctions such as visual/figural and episodic as well as acoustic memory. Although networking effects surely are involved in all memory subfunctions, the main brain target regions for verbal/episodic memory is the hippocampus (memory malfunctions are associated with hippocampal volume reduction and/or neuron losses) whereas those for other subfunctions are not known.

Therefore, morphological MBSR effects of the brain were compared to specific memory training via MBT. In this study, MBSR and MBT memory training are working as competitive effects on memory subfunctions, whereas a wellness massage and relaxing program and a do-not-change-anything group will serve as active and passive controls. The effects of memory function improvement by the respective training will be measured by MAT (Memory and Attention Test), a specific and validated computerized memory and attention test. Brain morphology was investigated by voxel based morphometry NMR before and immediately after an 8 weeks intervention period. Targets for morphometry are hippocampus CA1 region for verbal and episodic memory, the visual or acoustic cortex and the combined hippocampus areas for visual and acoustic memories, the amygdala volume for stress level and the frontotemporal lobe as a combined target of MBSR and memory assessment. Stress levels are measured by cortisol profiles of subjects. Compared were 4 groups- "MBSR" group- MBSR students after completed training, passive "control" group- subjects following an 8 weeks waiting period for the MBSR training without any memory training or wellness program, active control "MBT" group- subjects on an 8 week waiting period for the MBSR training doing an 8 week MBT memory training instead, "Wellness" group - doing a structured program using relaxing massage and calming computerized chair ("Brain Light").

The hypothesis of the study is that MBSR improves memory function better than MBT when measured by MAT. Compared to both active and passive controls, MBSR training induces specific morphologic changes in the brain, indicated by a volume change of the voxel based morphometry method of 5% of a defined brain region. In comparison to smaller and less neuroplasticity induced by MBT on memory brain regions, MBSR induces greater volume changes on hippocampus and amygdala and stress reduction than the wellness progam.

ELIGIBILITY:
Inclusion Criteria:

* willingness to do MBSR Training
* Age 25-65 years

Exclusion Criteria:

* history of ongoing or non-apparent psychosis under drug treatment
* drug addiction and intake
* non-willingness to accept the group allocation with the respective treatment
* non-compliance with a weekly trainings effort smaller than 20% of default

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Neuroplasticity | 8 weeks
  dose dependent changes in brain voxel based morphometry in NMR (volume reduction in %)

SECONDARY OUTCOMES:
well-being | 8 weeks
  dose dependent changes in well-being assessed with a standardized questionnaire (Score)
rumination | 8 weeks
  dose dependent changes in rumination assessed with a standardized questionnaire (score)
MAT | 8 weeks
  dose dependent changes in the computerized memory and attention test MAT (scores)
stress | 8 weeks
  dose dependent changes in individual cortisol levels (micrograms/liter)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Frietsch, MD, PhD, MBA, Study Chair — University Medicine Mannheim
Locations (1):
- Diakonissen Hospital, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No